CLINICAL TRIAL: NCT02886481
Title: Electrophysiologic Study of Perioperative Monitoring of the Recurrent Laryngeal Nerve: Impaired Vocal Cord Movement After Thyroidectomy
Acronym: NERLICORDE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2013_843_0013
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Recurrent Laryngeal Nerve
Keywords: thyroidectomy; Electrophysiologic; vocal cord movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: perioperative monitoring

SUMMARY:
Paralysis of the recurrent (or inferior) laryngeal nerve (RLN or ILN) is one of the most common and most serious complications of thyroid surgery. Neuromonitoring of the inferior laryngeal nerve (ILN or recurrent) is a technique currently used during thyroidectomy to locate ILN during dissection. Detector electrodes are placed in contact with vocal muscle which is stimulated electrically at the location of ILN, producing an acoustic and visual signal. This is a basic electromyographic technique whose diagnostic and prognostic potential for the entire neuromuscular system has not yet been fully explored. The study of action potentials generated by the stimulation-detection of nerves ILN and vagal nerves at the beginning and end of dissection, notably the decrease in amplitude, could allow a diagnosis during the course of surgery making it possible to diagnose lesions of the nerve and guide the surgeon in his surgical decisions, thus avoiding the risk of bilateral recurrent paralysis. It could also enable the surgeon to give a prognosis for functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a total thyroidectomy or a thyroid lobectomy

Exclusion Criteria:

* History of mobility disorder of the vocal cords

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a total thyroidectomy or a thyroid lobectomy
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
electrophysiologic state of the inferior laryngeal nerve | Day 1
  To study electrophysiologic state of the inferior laryngeal nerve with a neurostimulator during thyroidectomies in order to validate its diagnostic usefulness for ILN impairment of vocal cord movement.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir STRUNSKI, MD, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CHU Nimes, Nîmes